CLINICAL TRIAL: NCT04462536
Title: A Multicentre, Randomized, Double-blinded, Placebo-controlled, Parallel Group, Single-dose Design to Determine the Efficacy and Safety of Nerinetide in Participants With Acute Ischemic Stroke Undergoing Endovascular Thrombectomy Excluding Thrombolysis
Brief Title: Efficacy and Safety of Nerinetide in Participants With Acute Ischemic Stroke Undergoing Endovascular Thrombectomy Excluding Thrombolysis
Acronym: ESCAPE-NEXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NoNO Inc. (Industry)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA-1-009
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2023-09

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Vehicle only
  Interventions: Drug: Placebo
- Nerinetide (Experimental): Single intravenous infusion of nerinetide 2.6 mg/kg (up to a maximum dose of 270 mg) over 10 ± 1 minutes
  Interventions: Drug: Nerinetide

INTERVENTIONS:
Drug: Placebo — Vehicle only
  Arms: Placebo
Drug: Nerinetide — Single intravenous infusion of nerinetide 2.6 mg/kg (up to a maximum dose of 270 mg) over 10 ± 1 minutes
  Other Names: NA-1
  Arms: Nerinetide

SUMMARY:
The primary purpose of this study is to determine if a single dose of nerinetide can reduce global disability in people who have had a stroke and are selected for endovascular therapy without the use of a tissue plasminogen activator (alteplase, tenecteplase, or equivalent).

DETAILED DESCRIPTION:
This study is a Phase 3, randomized, multicentre, blinded, placebo-controlled, parallel group, single-dose with a single interim analysis. Because AIS (acute ischemic stroke) is a medical emergency, the trial is designed to enable the administration of standard-of-care treatments without delay in order to save the life of the person concerned, restore good health or alleviate suffering.

Participants harboring an acute ischemic stroke who are selected for endovascular revascularization without intravenous or intra-arterial thrombolytic therapy will be given a single, 2.6 mg/kg (up to a maximum dose of 270 mg) intravenous dose of nerinetide or placebo. Outcomes of the main trial will be evaluated throughout a 90 day observation period.

Participants will be followed at 1-Year for the analytic sub-trial for further outcome assessment by telemedicine or telephone interview conducted by individuals blinded to the outcome of the main trial. This sub-trial will be conducted to explore the independent functioning and quality of life at 1-Year.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke (AIS) selected for emergency endovascular treatment.
2. Age 18 years or greater.
3. Onset (last-known-well) time to randomization time within 12 hours.
4. Disabling stroke defined as a baseline National Institutes of Health Stroke Score (NIHSS):

   1. NIHSS > 5 for internal carotid artery (ICA) and M1-middle cerebral artery (MCA) occlusion; or
   2. NIHSS > 10 for M2-MCA occlusion.
5. Confirmed symptomatic intracranial occlusion at one or more of the following locations: Intracranial carotid I/T/L, M1 or M2 segment MCA. Tandem extracranial carotid and intracranial occlusions are permitted.
6. Pre-stroke (24 hours prior to stroke onset) independent functional status in activities of daily living with modified Barthel Index (BI) ≥ 95. Patient must be living without requiring nursing care.
7. Qualifying imaging performed less than 2 hours prior to randomization.
8. Consent process completed as per national laws and regulation and the applicable ethics committee requirements.

Exclusion Criteria:

1. Treated with a tissue plasminogen activator (e.g., alteplase or tenecteplase) within 24 hours before randomization.
2. Determination by the treating physician, based on current treatment guidelines and medical evidence, that treatment with a plasminogen activator is indicated.
3. Large core of established infarction defined as ASPECTS 0-4.
4. Absent or poor collateral circulation on qualifying imaging (e.g. collateral score of 0 or 1).
5. Any intracranial hemorrhage on the qualifying imaging.
6. Planned use of an endovascular device not having approval or clearance by the relevant regulatory authority.
7. Endovascular thrombectomy procedure is completed as defined by the presence of TICI 2c/3 reperfusion or completion of groin / arterial closure.
8. Clinical history, past imaging or clinical judgment suggesting that the intracranial occlusion is chronic or there is suspected intracranial dissection such that there is a predicted lack of success with endovascular intervention.
9. Estimated or known weight > 120 kg (264 lbs).
10. Pregnancy/Lactation; female, with positive urine or serum beta human chorionic gonadotropin (β-hCG) test, or breastfeeding.
11. Known prior receipt of nerinetide for any reason, including prior enrolment in this ESCAPE-NEXT trial.
12. Severe known renal impairment defined as requiring renal replacement therapy (hemo- or peritoneal dialysis).
13. Severe or fatal comorbid illness that will prevent improvement or follow up.
14. Inability to complete follow-up treatment to Day 90.
15. Participation in another clinical trial investigating a drug, medical device, or a medical procedure in the 30 days preceding trial inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Hill, MD MSc, Principal Investigator — Study Principal Investigator, University of Calgary
Locations (81):
- United States (17):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Providence Little Company of Mary Medical Center - Torrance, Torrance, California
  - Swedish Medical Center, Englewood, Colorado
  - Baptist Health Research Institute, Jacksonville, Florida
  - University of Miami, Jackson Memorial Hospital, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - NYU Langone Hospital Brooklyn, Brooklyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Ohio State University, Wexner Medical Center Neurological Surgery, Columbus, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC Stroke Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Valley Baptist Medical Center - Harlingen, Harlingen, Texas
  - Swedish Medical Center - Cherry Hill Campus, Seattle, Washington
- Australia (8):
  - Royal Adelaide Hospital, Adelaide
  - Princess Alexandra Hospital, Brisbane
  - Monash Medical Centre, Clayton
  - Gold Coast University Hospital, Gold Coast
  - Fiona Stanley Hospital, Murdoch
  - Sir Charles Gairdner Hospital, Nedlands
  - John Hunter Hospital, Newcastle
  - Royal Melbourne Hospital, Parkville
- Canada (16):
  - Foothills Medical Centre - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre (LHSC), London, Ontario
  - Ottawa Hospital Research Institute (OHRI), Ottawa, Ontario
  - St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - University Hospital of Montreal, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Germany (23):
  - Universitätsklinikum RWTH Aachen, Aachen
  - Klinikum Altenburger Land GmbH, Altenburg
  - Universitätsklinikum Augsburg, Augsburg
  - Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Dortmund gGmbH, Dortmund
  - University of Dresden, Dresden
  - Alfried-Krupp-Krankenhaus, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Göttingen University Hospital, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Heidelberg University Hospital, Heidelberg
  - University Hospital Schleswig-Holstein, Kiel
  - Universitätsklinikum Leipzig - Klinik und Poliklinik für Neurologie, Leipzig
  - Klinikum rechts der Isar Technical University of Munich, München
  - LMU Klinikum München, München
  - Universitätsklinikum Münster, Münster
  - Nürnberg Hospital South Campus, Nuremberg
  - Evangelisches Krankenhaus Oldenburg, Oldenburg
  - Klinikum Stuttgart, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Würzburg University Hospital, Würzburg
- Italy (5):
  - Ospedale Maggiore di Bologna "Carlo Alberto Pizzardi", Bologna
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino, Genoa
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Antonio Cardarelli, Napoli
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Maastricht University Medical Center, Maastricht
  - Erasmus University Medical Center, Rotterdam
- Norway (4):
  - Oslo University Hospital Rikshospitalet, Oslo
  - Oslo University Hospital Ulleval, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North-Norway, Tromsø
- Singapore (2):
  - National Neuroscience Institute, Singapore
  - National University Hospital, Singapore
- Switzerland (3):
  - Kantonsspital Aarau, Aarau
  - Universitätsspital Basel, Basel
  - Universitatsklinik fur Neurologie, Inselspital, Bern

REFERENCES:
- [Derived] Hill MD, Goyal M, Demchuk AM, Menon BK, Field TS, Guest WC, Berrouschot J, Bormann A, Pham M, Haeusler KG, Dippel DWJ, van Doormaal PJ, Dorn F, Bode FJ, van Adel BA, Sahlas DJ, Swartz RH, Da Costa L, Ospel JM, McDonough RV, Ryckborst KJ, Almekhlafi MA, Heard KJ, Garman DJ, Adams C, Kohli Y, Schoon BA, Buck BH, Muto M, Zafar A, Schneider H, Grossberg JA, Yeo LLL, Tarpley JW, Psychogios MN, Coutinho JM, Limbucci N, Puetz V, Kelly ME, Campbell BCV, Poli S, Poppe AY, Shankar JJ, Chandra R, Dowlatshahi D, Lopez GA, Cirillo L, Moussaddy A, Devlin M, Garcia-Bermejo P, Mandzia JL, Skjelland M, Aamodt AH, Silver FL, Kleinig TJ, Pero G, Minnerup J, McTaggart RA, Puri AS, Chiu AHY, Reimann G, Gubitz GJ, Camden MC, Lee SK, Sauvageau E, Mundiyanapurath S, Frei DF, Choe H, Rocha M, Gralla J, Bailey P, Fischer S, Liebig T, Dimitriadis K, Gandhi D, Chapot R, Jin A, Hassan AE, Zwam WV, Maier IL, Wiesmann M, Niesen WD, Advani R, Eltoft A, Asdaghi N, Murphy C, Remonda L, Ghia D, Jansen O, Holtmannspoetter M, Hellstern V, Witt K, Fromme A, Nimjee SM, Turkel-Parella D, Michalski D, Maegerlein C, Tham CH, Tymianski M; ESCAPE-NEXT Investigators. Efficacy and safety of nerinetide in acute ischaemic stroke in patients undergoing endovascular thrombectomy without previous thrombolysis (ESCAPE-NEXT): a multicentre, double-blind, randomised controlled trial. Lancet. 2025 Feb 15;405(10478):560-570. doi: 10.1016/S0140-6736(25)00194-1. PMID 39955119

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Nerinetide
Started | 396 | 454
Received Study Medication | 393 | 451
Completed | 391 | 441
Not Completed | 5 | 13
Not completed — Withdrawal by Subject | 3 | 9
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nerinetide | Total
Number analyzed (Participants) | 393 | 451 | 844
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 102 | 196
  >=65 years | 299 | 349 | 648
Age, Continuous [Median (Standard Deviation); unit: years] | 75 (12.56) | 76 (13.29) | 76 (12.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 223 | 417
  Male | 199 | 228 | 427
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 38 | 62
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
  Black or African American | 13 | 18 | 31
  White | 323 | 362 | 685
  More than one race | 15 | 21 | 36
  Unknown or Not Reported | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Independent Functioning on the Modified Rankin Scale (mRS), as Defined by a Score of 0-2
Description: The modified Rankin Scale (mRS) is a valid and reliable clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke. It is a scale used to measure functional recovery (the degree of disability or dependence in daily activities) of people who have suffered a stroke. mRS scores range from 0 (best outcome) to 6 (worst outcome), with 0 indicating no residual symptoms; 5 indicating bedbound, requiring constant care; and 6 indicating death.
Time Frame: 90 days
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide
Number analyzed (Participants) | 396 | 454
Participants | 181 | 206

2. Secondary Outcome: Mortality Rate, as Defined by Event Rate (Percent) for Mortality Over the 90-day Study Period.
Description: The estimand of mortality rate was the adjusted unconditional population difference in the number of deaths observed divided by the number of participants observed over the 90-day study period (mortality proportions) between treatment conditions (nerinetide vs. placebo) in the target patient population at Day 90. Deaths occurring over the Day 90 period were considered as non-responses.
Time Frame: 90 days
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide
Number analyzed (Participants) | 396 | 454
Participants | 70 | 87

3. Secondary Outcome: Number of Participants Exhibiting a Worsening of Their Index Stroke.
Description: Worsening of stroke is defined as (A) progression, or hemorrhagic transformation of the index stroke, as documented by medical imaging that is (a) life-threatening requiring intervention and/or (b) results in increased disability as gauged by a ≥4 point increase from lowest NIHSS during hospitalization or (B) results in death from the index stroke.
Time Frame: 90 days
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide
Number analyzed (Participants) | 396 | 454
Participants | 68 | 76

4. Secondary Outcome: Number of Participants With Good Neurological Outcome, as Defined by a Score of 0-2 on the NIHSS at Day 90 Post Randomization.
Description: The National Institutes of Health Stroke Scale (NIHSS) is a standardized neurological examination score that is a valid and reliable measure of disability and recovery after acute stroke. Scores range from 0 to 42, with higher scores indicating increasing severity.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide
Number analyzed (Participants) | 396 | 454
Participants | 251 | 268

ADVERSE EVENTS:
Time Frame: TEAEs occurring within 30 days of randomization and all SAEs up to the end of study visit (Day 90 visit or death)
Arm/Group | Placebo | Nerinetide
All-Cause Mortality (participants affected / at risk) | 70/396 | 87/454
Serious Adverse Events (participants affected / at risk) | 148/393 | 182/451
Other Adverse Events (participants affected / at risk) | 329/393 | 393/451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=393) | Nerinetide (N=451)
Stroke in Evolution (Nervous system disorders) | 35 | 29
ischaemic stroke (Nervous system disorders) | 14 | 22
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Haemorrhagic transformation stroke (Nervous system disorders) | 3 | 8
Cerebral haemorrhage (Nervous system disorders) | 3 | 8
Pneumonia (Infections and infestations) | 7 | 8
Cardiac failure congestive (Cardiac disorders) | 3 | 8
Atrial fibrillation (Cardiac disorders) | 2 | 7
Failure to thrive (Metabolism and nutrition disorders) | 7 | 8
various - combined (Vascular disorders) | 10 | 8
various-combined (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 11
various - combined (Injury, poisoning and procedural complications) | 5 | 10
various-combined (Psychiatric disorders) | 9 | 5
various - combined (General disorders) | 3 | 7
various (Renal and urinary disorders) | 7 | 3
others - combined (Nervous system disorders) | 19 | 31
others - combined (Infections and infestations) | 18 | 24
others -combined (Respiratory, thoracic and mediastinal disorders) | 12 | 18
others-combined (Cardiac disorders) | 13 | 16
others-combined (Metabolism and nutrition disorders) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=393) | Nerinetide (N=451)
Urinary Tract infection (Infections and infestations) | 46 | 52
Hypotension (Vascular disorders) | 36 | 54
Haemorrhagic transformation stroke (Nervous system disorders) | 39 | 50
Headache (Nervous system disorders) | 26 | 52
Hypokalaemia (Metabolism and nutrition disorders) | 34 | 47
pyrexia (General disorders) | 36 | 35
Pneumonia aspriation (Respiratory, thoracic and mediastinal disorders) | 18 | 24
constipation (Gastrointestinal disorders) | 20 | 36
Atrial fibrillation (Cardiac disorders) | 15 | 22
Pneumonia (Infections and infestations) | 20 | 13
Delirium (Psychiatric disorders) | 21 | 21
Bradycardia (Cardiac disorders) | 18 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04462536/Prot_SAP_000.pdf